CLINICAL TRIAL: NCT06016634
Title: A Feasibility Study of Alendronate as Treatment for Osteonecrosis in Adults With Sickle Cell Disease
Brief Title: Alendronate for Osteonecrosis in Adults With Sickle Cell Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1693339; 5K23HL148310 (NIH); 2020095 (Other Grant/Funding Number: Doris Duke Charitable Foundation)
Record Dates: First submitted 2023-08-07; First posted 2023-08-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Osteonecrosis; Ischemic Necrosis; Avascular Necrosis
Keywords: sickle cell disease; sickle cell anemia; osteonecrosis of the femoral head; hip osteonecrosis; ischemic necrosis of the femur; avascular necrosis of the femur
MeSH Terms: conditions — Anemia, Sickle Cell; Osteonecrosis; Legg-Calve-Perthes Disease | interventions — Alendronate

STUDY DESIGN:
Intervention Model Description: Prospective cohort of 30 adults with sickle cell disease and hip osteonecrosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alendronate group (Experimental): Single-arm prospective cohort of 30 adult with SCD
  Interventions: Drug: Alendronate Sodium

INTERVENTIONS:
Drug: Alendronate Sodium — Administer oral alendronate 70 mg once a week x 24 weeks to all study participants
  Other Names: alendronate tablet; oral alendronate; Fosamax; Binosto

SUMMARY:
A prospective, single-arm, intervention study of oral alendronate in adults with sickle cell disease and osteonecrosis

DETAILED DESCRIPTION:
The investigators hypothesize that adults with sickle cell disease (SCD) and osteonecrosis of the femoral (hip) and/or humeral (shoulder) heads will tolerate oral alendronate 70 mg administered once a week x 24 weeks (6 months). In addition to collecting safety and tolerability data on alendronate in study participants, the investigators will also measure the preliminary efficacy of alendronate using changes in the Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) Pain Impact scores from baseline to 3-months and 6-months after alendronate initiation. Serum and urine specimen will also be collected to assess changes in bone biomarkers at baseline, 3-months, and 6-months.

The investigators plan to recruit 24 adults with SCD from the University of California Davis Medical Center to this single-arm, open label, interventional study. The investigators anticipate enrolling 1-2 participants per month between Sep 2024- Dec 2025.

The study endpoints are summarized below:

* To determine the recruitment and retention rates of adults with SCD and osteonecrosis enrolled in this prospective, single-arm, open label alendronate interventional study
* To measure the safety, tolerability, and preliminary efficacy of oral alendronate in adults with SCD-related osteonecrosis over a 6-month treatment duration
* To measure changes in bone biomarkers in the serum and urine of study participants not receiving chronic red blood cell transfusions at 3 time points: baseline, 3-months, and 6-months after initiation of alendronate

The investigators' goal is to complete primary data analysis by May 2026.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years with SCD (any genotype, confirmed by hemoglobin electrophoresis or high performance liquid chromatography)
* Ability to provide written informed consent
* Ability to lay on a dual-energy X-ray absorptiometry (DXA) scanner
* Negative urine pregnancy test for anyone of childbearing potential at study entry

Exclusion Criteria:

* Pregnant women
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Hospitalizations (for any cause) within 2 weeks of study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | up to 28 weeks
  Proportion of eligible patients who get recruited to the study; number of enrolled patients who complete 6-month study
Incidence of Treatment-Emergent Adverse Events as assessed by participant report | up to 28 weeks
  Collect all adverse events reported by patients and determine if related to study drug
Pain assessed by the Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) Pain Impact questionnaire | up to 28 weeks
  The Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) Pain Impact questionnaire is a patient-reported outcome measure of pain level in the past 7 days. The ASCQ-Me pain scale ranges from 0-100, with a standardized mean of 50 and a standard deviation of 10, where lower scores signify worse disease impact.

SECONDARY OUTCOMES:
Serum CTX-1 | baseline, 3 months, 6 months
  Measurement of C-terminal telopeptide of type I collagen (CTX) in serum as a biomarker for osteoclast activity (bone resorption)
Serum P1NP | baseline, 3 months, 6 months
  Measurement of Procollagen type I N-terminal propeptide (P1NP) in serum as a biomarker for osteoblast activity (bone formation)

CONTACTS AND LOCATIONS:
Overall Officials: Oyebimpe O Adesina, MD, MS, Principal Investigator — UC Davis School of Medicine
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No